CLINICAL TRIAL: NCT03781999
Title: The Effect of a Combination of Orange- and Pomegranate Actives on Physical Fitness in Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioActor (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Actiful_001
Record Dates: First submitted 2018-12-10; First posted 2018-12-20 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Fitness
Keywords: Performance; Polyphenols; Nutrition; Sports

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Actiful (Experimental): a supplement containing 500 mg orange extract and 200 mg pomegranate actives
  Interventions: Dietary Supplement: Actiful
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Actiful — supplement containing 500 mg orange extract and 200 mg pomegranate actives
  Arms: Actiful
Other: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the effect of daily supplementation of a combined orange- and pomegranate extract for a period of 4 weeks on physical fitness compared to placebo.

In this crossover study, participants will daily receive either a placebo or Actiful®, a supplement containing 500 mg orange extract and 200 mg pomegranate actives, for 4 weeks followed by a wash-out period of 4 to 8 weeks. Subsequently, the second intervention period of 4 weeks (active product or placebo) will take place. The product and placebo will be supplied in capsules that participants can ingest with a glas of water (daily, prior to breakfast).

DETAILED DESCRIPTION:
Dietary habits and physical activity are two important components of a healthy lifestyle. Targeted nutritional interventions may improve health and stimulate physical activity. Both orange extracts and pomegranate concentrate have been shown to exert beneficial effects on health and exercise performance. However, the effects of a combination of the two extracts on exercise and physical activity have not been investigated yet. It is expected that this combination may be an effective dietary way to improve exercise performance, physical activity in the free-living state, and quality of life in a middle aged population.

ELIGIBILITY:
Inclusion Criteria:

* 60 - 75 years old
* non smoking
* BMI 18 -28 kg/m²

Exclusion Criteria:

* Allergy to test product/placebo or citrus fruits
* BMI lower than 18 or higher than 28
* Recent muscle injury in less than one month before the start of the study
* Inability to perform the fitness tests
* Medical conditions that might influence outcome measure or participant safety during testing, including but not limited to: severe cardiovascular disease, cancer, Parkinson's disease. To be decided by PI.
* High blood pressure (systolic ≥ 140 mmHg, diastolic ≥ 90 mmHg)
* Use of medication that may interfere with the study results, use of beta-blockers
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study
* Abuse of products; alcohol (> 20 alcoholic units per week) and drugs

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
6 Minute Walking Test | 0-4-8-12 weeks
  Participants have to walk for 6 minutes, as fast as possible. Total distance will be measured.

SECONDARY OUTCOMES:
Senior Fitness test | 0-4-8-12 weeks
  Fitness tests to see if Actiful improves physical activity level
Daily physical activity measured by accelerometers | 0-4-8-12 weeks
  Accelerometer is worn for 7 days prior to each testing day
Quality of life questionnaire - WHOQOL-100 | 0-4-8-12 weeks
  Participants will be asked to fill out the WHOQOL-100 questionnaire to determine quality of life. Scale from 1-5 (disagree-agree)
Concentration of blood marker TAC | 0-4-8-12 weeks
  Total antioxidant capacity measurement in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Troost, Dr, Principal Investigator — Maastricht University
Locations (1):
- BioActor, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bednarska K, Fecka I, Scheijen JLJM, Ahles S, Vangrieken P, Schalkwijk CG. A Citrus and Pomegranate Complex Reduces Methylglyoxal in Healthy Elderly Subjects: Secondary Analysis of a Double-Blind Randomized Cross-Over Clinical Trial. Int J Mol Sci. 2023 Aug 24;24(17):13168. doi: 10.3390/ijms241713168. PMID 37685975